CLINICAL TRIAL: NCT02202954
Title: Comparison of Two Rehabilitation Strategies in Patients With Hemiparesis One Year or More After Stroke. Efficacy and Cost After One Year Treatment. A Randomized, Controlled, Multicenter, Single Blind Study
Brief Title: Comparison of Two Rehabilitation Strategies in Patients With Hemiparesis One Year or More After Stroke
Acronym: NEURORESTORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P100114; 2012-A00348-35 (Other: ID RCB)
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Hemiparesis
Keywords: Stroke; Muscle Spasticity; Rehabilitation
MeSH Terms: conditions — Paresis; Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guided Self-rehabilitation Contract (Active Comparator): In Guided Self-rehabilitation Contracts, the therapist acts as a coach, in the sports' sense, providing double guidance: technical, selecting and teaching the required exercises to the patient using infrequent thorough visits, for example every month; Psychological, binding with the patient on the contract.
  The patient agrees to perform the prescribed daily stretch postures and rapid alternating movements over the long term and to document this work in a written diary.
  Interventions: Other: Guided Self-rehabilitation Contract
- Conventional rehabilitation (No Intervention): conventional therapy in the community

INTERVENTIONS:
Other: Guided Self-rehabilitation Contract — In Guided Self-rehabilitation Contracts, the therapist acts as a coach, in the sports' sense, providing double guidance: technical, selecting and teaching the required exercises to the patient using infrequent thorough visits, for example every month; Psychological, binding with the patient on the contract.
  The patient agrees to perform the prescribed daily stretch postures and rapid alternating movements over the long term and to document this work in a written diary.
  Arms: Guided Self-rehabilitation Contract

SUMMARY:
In the situation of motor limitations that people often experience after stroke, current health systems cannot provide for the daily amount and duration of high intensity muscle stretch and motor training that would be required over protracted periods to involve muscle and brain plasticity. For patients with sufficient cognitive abilities, Guided Self-rehabilitation Contracts allow implementing stretch and training at high intensity and may result in meaningful functional improvement in chronic stages, as long as discipline persists over at least a year span.

This single blind control protocol will evaluate Guided Self-rehabilitation Contracts as against conventional therapy in the community, for a one year duration in persons with chronic hemiparesis after stroke.

DETAILED DESCRIPTION:
This single blind controlled multicentre protocol will compare the evolution after a one-year treatment, either using a Guided Self-rehabilitation Contract or conventional therapy in the community. Patients with chronic stroke-induced hemiparesis (over a year post stroke) will be selected to be randomized between the two groups, Conventional or in Guided Self-rehabilitation Contracts.

In Guided Self-rehabilitation Contracts, the therapist acts as a coach, in the sports' sense, providing double guidance:

* Technical, selecting and teaching the required exercises to the patient using infrequent thorough visits, for example every month.
* Psychological, binding with the patient on the contract.

The patient agrees to:

* Perform the prescribed daily stretch postures and rapid alternating movements over the long term.
* Document this work in a written diary.

To facilitate such contracts, a manual for guided self-rehabilitation in spastic paresis has been developed and will be provided to patients randomized to that group.

124 patients will be enrolled from 6 centers in France: Creteil, Paris Fernand-Widal, Toulouse, Reims, Saint-Etienne and Bordeaux. The duration of patient participation will be 2 years: 6 months follow-up, 1 year intervention and another 6-month follow-up after the study intervention. Only functional assessments will be used, using in particular ambulation speed for the lower limb and the Modified FRENCHAY Scale for the upper limb.

ELIGIBILITY:
Inclusion Criteria:

* Patient with spastic hemiparesis, following a unique stroke episode over a year before enrollment into the study
* Age ≥ 18
* Barefoot walking possible with no assistive device over 10 m
* Fast barefoot ambulation speed between 0.1 m/sec and 1.3 m/sec
* Mean Modified FRENCHAY Score between 2 and 8/10
* Patient having provided a signed consent to participate in this trial

Exclusion Criteria:

* Multiple stroke episodes, clinically of based on brain imaging
* No recent (less than 3 months before enrollment) brain imaging (CT scan or MRI) in case of doubt about multiple stroke episodes
* Concurrent severe condition jeopardizing functional or vital prognosis, or the ability to participate in rehabilitation sessions
* Cognitive, phasic or behavioral condition impeding verbal communication, active participation to a rehabilitation or self-rehabilitation program, or participation in a research study, according to the investigator's judgment
* Person having a tutor or benefiting from a law protection order
* Person not benefiting from French State Health Insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Functional motor recovery assessed by a composite endpoint (one for upper limbs and one for lower limbs) | After one year of treatment
  1. Fast 10-meter barefoot ambulation speed with no assistive device
  2. Active upper limb function using the Modified FRENCHAY scale (10 everyday life activities performed live in front of the investigator and videotaped - videos reviewed later by a blinded investigator).

SECONDARY OUTCOMES:
Speed, step length and cadence over 10 meters at comfortable speed, barefoot and with shoes, with no assistive device | One assessment visit every 6 month for 2 years
Speed, step length, cadence and physiological cost index over 2 minutes at maximal speed, with shoes | One assessment visit every 6 month for 2 years
Disability Assessment Scale: interview between patient and investigator, assessing the level of disability in 4 domains (dressing, cosmesis, hygiene and pain) | One assessment visit every 6 month for 2 years
Barthel Activity of Daily Living (ADL) Index | One assessment visit every 6 month for 2 years
Euro-Qol - 5 dimension (EQ-5D) | One assessment visit every 6 month for 2 years
  European Quality of Life Scale
Geriatric Depression Scale - 15 | One assessment visit every 6 month for 2 years
Questionnaire to the patient (or caregiver) evaluating monthly frequency of physical therapy sessions and amount of home aid during the whole study period, that will serve as basis for a cost evaluation from the point of view of medical insurance. | One assessment visit every 6 month for 2 years
Estimation of the total cost of care, including medical costs, social expenses, amount of social benefits, from the point of view of the medical insurance and of the state, to include all payors. | One assessment visit every 6 month for 2 years

OTHER OUTCOMES:
Evaluation by the occupational therapist of home adaptation and the functioning at home | One assessment visit every 6 month for 2 years
  An ancillary study on the 44 patients in the Paris area
Evaluation by a clinical psychologist of coping with each type of care (guided self-rehabilitation or conventional), of the required psychological resources and the potential need for psychological follow-up. | One assessment visit every 6 month for 2 years
  An ancillary study on the 44 patients in the Paris area.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel GRACIES, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Derived] Gracies JM, Pradines M, Ghedira M, Loche CM, Mardale V, Hennegrave C, Gault-Colas C, Audureau E, Hutin E, Baude M, Bayle N; Neurorestore Study Group. Guided Self-rehabilitation Contract vs conventional therapy in chronic stroke-induced hemiparesis: NEURORESTORE, a multicenter randomized controlled trial. BMC Neurol. 2019 Mar 12;19(1):39. doi: 10.1186/s12883-019-1257-y. PMID 30871480